CLINICAL TRIAL: NCT06920316
Title: Digital Diet and Exercise Intervention to Reduce Liver Fibrosis in Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD): A Pilot Randomised Controlled Trial
Brief Title: Digital Diet and Exercise Intervention to Reduce Liver Fibrosis in Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD)
Acronym: DEFIB-MASLD
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: St. George's Hospital, London (Other)
Responsible Party: Principal Investigator, Caroline Gosson, Principal Investigator, Hepatology Clinical Research Fellow, St. George's Hospital, London
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: StGeorgesLondon
Record Dates: First submitted 2025-01-29; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Non-alcoholic Fatty Liver Disease; Fatty liver; Digital health
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gro Health Application (Active Comparator): The Gro Health digital application is a personalised treatment platform proven to support sustainable weight loss. It is non-MHRA regulated as MASLD is within the device's UKCA/CE UKNI/CE marked indication. Gro Health reports 7% weight loss at 52 weeks in patients with Type 2 Diabetes Mellitus. We can set up the application so patients follow a Mediterranean diet. Over 1000 recipes of different cuisines will be available, along with weekly diet plans and shopping lists. Based on the patient's body mass index, daily calories and macronutrient targets will be calculated in line with the Mediterranean diet. Aerobic exercise can be tracked by daily step count linked by compatible smartwatches and smartphones. Physical activity can also be logged manually. Gro Health provides educational videos on aerobic and resistance exercise, along with 'follow along' videos of exercises for patients. These videos range from ones for beginners to those who have more experience with exercise.
  Interventions: Device: Gro Health digital application
- Standard of Care (No Intervention): If randomised to this arm, participants will not receiving any additional intervention beyond their usual clinical care for their condition.

INTERVENTIONS:
Device: Gro Health digital application — The Gro Health digital application is a personalised treatment platform proven to support sustainable weight loss. It is non-MHRA regulated as MASLD is within the device's UKCA/CE UKNI/CE marked indication. Gro Health reports 7% weight loss at 52 weeks in patients with Type 2 Diabetes Mellitus. We can set up the application so patients follow a Mediterranean diet. Over 1000 recipes of different cuisines will be available, along with weekly diet plans and shopping lists. Based on the patient's body mass index, daily calories and macronutrient targets will be calculated in line with the Mediterranean diet. Aerobic exercise can be tracked by daily step count linked by compatible smartwatches and smartphones. Physical activity can also be logged manually. Gro Health provides educational videos on aerobic and resistance exercise, along with 'follow along' videos of exercises for patients. These videos range from ones for beginners to those who have more experience with exercise.
  Arms: Gro Health Application

SUMMARY:
Study Title: Digital Diet and Exercise Intervention to Reduce Liver Fibrosis in Metabolic Dysfunction-associated Steatotic Liver Disease (MASLD): A Randomized Controlled Trial (D-FIB-MASLD)

Objective:

This study aims to assess whether a digital application called Gro Health can help patients with MASLD and significant liver fibrosis reduce their liver stiffness. Liver stiffness is a measure of liver health and fibrosis. The study will also investigate the impact of this intervention on weight, body measurements, liver health markers, and overall quality of life.

Background:

MASLD is a liver condition linked to metabolic issues such as obesity and diabetes. It is a common cause of liver-related complications and can lead to severe liver damage. Lifestyle changes, like improved diet and exercise, are key to managing MASLD, but achieving these changes can be challenging for many patients. Digital tools like the Gro Health app may provide personalized and accessible support to improve outcomes.

Study Design:

This is a randomized controlled trial involving 100 participants with MASLD and significant fibrosis. Participants will be assigned to either the intervention group (using the Gro Health app) or a control group (receiving standard care). The study will take place at a single site over 12 months.

Intervention:

Participants in the intervention group will use the Gro Health app, which offers personalized calorie and activity goals, a food diary, over 1,000 Mediterranean diet recipes, and educational resources. They will also receive a smartwatch to track steps and physical activity. The app includes a feature allowing researchers to monitor participants' engagement and provide encouragement.

Eligibility:

Adults aged 18 or older with a diagnosis of MASLD and a liver stiffness measurement of 8 kPa or higher are eligible. Key exclusions include alcohol consumption over 14 units/week, a BMI over 40, or certain other liver diseases or medications.

Outcomes:

The primary outcome is a reduction in liver stiffness after six months. Secondary outcomes include changes in weight, BMI, body fat percentage, liver enzymes, cholesterol, and quality of life. Additional data on app usage, physical activity, and dietary habits will also be collected for the intervention group.

Potential Impact:

If successful, this study will provide evidence that digital tools can help improve liver health and overall well-being in patients with MASLD, offering a scalable solution for healthcare systems.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and over
* Diagnosis of MASLD made by a hepatologist
* Vibration-Controlled Transient Elastography (VCTE) (FibroScan) liver stiffness measurement (LSM) 8 kPa and above
* Able to provide written consent
* Own a smartphone with data plan

Exclusion Criteria:

* Alcohol consumption >14 units/week
* BMI >40
* Liver disease due to: Alcohol including MASLD with increased alcohol intake (MetALD), Any viral hepatitis, Autoimmune and cholestatic aetiologies including, but not limited to, primary biliary cholangitis and primary sclerosing cholangitis, Hereditary aetiologies including, but not limited to, haemachromatosis, Wilson's disease, alpha-1-antitrypsin deficiency
* Currently under investigation for cancer or receiving treatment for active cancer
* Myocardial infarction within last 6 months or uncontrolled cardiovascular disease
* Pregnant or planning
* Currently or due to be taking any of the following drugs: GLP-1/GIP agonists, Systemic high dose corticosteroids for >6 weeks, Tamoxifen, Amiodarone, Methotrexate, Lomitapide, Valproate, Irinotecan, 5-Fluoruracil
* Currently using or enrolled in any other lifestyle intervention application or weight loss programme
* Undergone or due to undergo bariatric surgery including bariatric endoscopic procedures
* Any other intercurrent illness that is either life-threatening or of clinical significance such that it might limit compliance with study procedures, in the Investigator's opinion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is change in liver stiffness measurement at 6 months compared to baseline | 6 months
  The primary outcome measure is change in liver stiffness measurement (LSM) at 6 months compared to baseline. LSM is measured in kPa.
  Vibration controlled transient elastography (VCTE) has been validated as a measure of fibrosis across a wide spectrum of chronic liver diseases including MASLD. Whilst liver histology remains the gold standard for fibrosis staging, and magnetic resonance imaging and elastography for non-invasive hepatic lipid quantification and fibrosis respectively, both techniques are largely limited by being time consuming and expensive. VCTE provides multiple advantages of low cost, short procedure time, immediate result availability, good reproducibility and the ability to be performed in an outpatient setting.
  Studies have shown that LSM has good accuracy for liver-related events and mortality. Change in LSM has been shown to correlate with the risk of liver-related events and death.

SECONDARY OUTCOMES:
Weight in kilograms - To compare the effect of a digital application based lifestyle intervention to standard of care on weight | 6 and 12 months
  Baseline weight in kilograms will be taken at day 0 on calibrated hospital scales in clinic from all study participants. A formal weight will be taken at all hospital clinic appointments and at 26 weeks and at the end of the intervention period. Only weights taken on the calibrated hospital scales will be used for analysis.
Percentage weight loss - To compare the effect of a digital application based lifestyle intervention to standard of care on percentage weight loss | 6 and 12 months
  Baseline weight in kilograms will be taken at day 0 on calibrated hospital scales in clinic from all study participants. A formal weight will be taken at all hospital clinic appointments and at 26 weeks and at the end of the intervention period. Only weights taken on the calibrated hospital scales will be used for analysis.
Height in metres | baseline
  Height in metres will be taken at baseline for the use in BMI calculation as stated for BMI outcome
Body mass index - To compare the effect of a digital application based lifestyle intervention to standard of care on BMI | 6 and 12 months
  Baseline weight in kilograms will be taken at day 0 on calibrated hospital scales in clinic from all study participants. Baseline height will be taken at day 0 only. A formal weight will be taken at all hospital clinic appointments and at 26 weeks and at the end of the intervention period. Only weights taken on the calibrated hospital scales will be used for analysis.
Body fat percentage - To compare the effect of a digital application based lifestyle intervention to standard of care on body fat percentage | 6 and 12 months
  Measured at baseline, 26 weeks and at the end of the intervention period using Withings smart scale
Controlled Attenuation Parameter - To compare the effect of a digital application based lifestyle intervention to standard of care on CAP. | 6 and 12 months
  CAP is a measure of liver fat taken by Vibration Controlled Transient Elastography (also known as Fibroscan). Baseline CAP will be taken on day 0 using FibroScan machine by a trained operator who is not involved in the trial from all study participants. A reading will be taken at 26 weeks and at the end of the intervention period.
Spleen stiffness measurement - To compare the effect of a digital application based lifestyle intervention to standard of care on SSM | 6 and 12 months
  Spleen stiffness measurement is measured by vibration controlled transient elastography (also known as Fibroscan) and indicates spleen scarring. Baseline SSM will be taken on day 0 using FibroScan machine by a trained operator who is not involved in the trial from all study participants. A reading will be taken at 26 weeks and at the end of the intervention period.
To compare the effect of a digital application based lifestyle intervention to standard of care on the following blood parameters: alanine transaminase ALT, aspartate aminotransferase AST, HbA1c | 6 and 12 months
  Concentration of ALT, AST, HbA1c in blood samples will be taken on day 0, 26 weeks and at the end of the intervention period from all participants if not taken within the last 3 months
To compare the effect of a digital application based lifestyle intervention to standard of care on the following blood parameters: total cholesterol, low-density lipoprotein cholesterol LDL, high-density lipoprotein cholesterol HDL, triglycerides | 6 and 12 months
  Concentration of total cholesterol, LDL, HDL and triglycerides in blood samples will be taken on day 0, 26 weeks and at the end of the intervention period from all participants if not taken within the last 3 months.
Waist and hip circumference - To compare the effect of a digital application based lifestyle intervention to standard of care on these measurements | 6 and 12 months
  Baseline waist and hip circumference will be measured on day 0 using a tape measure in centimetres at the midpoint between the lower margin of the last palpable rib and the top of the iliac crest as recommended by the WHO from all study participants. A measurement will be taken at 26 weeks and at the end of the intervention period.
Systolic blood pressure - To compare the effect of a digital application based lifestyle intervention to standard of care on blood pressure | 6 and 12 months
  Baseline systolic blood pressure will be taken on day 0 from all study participants. A reading will be taken at 26 weeks and the end of the intervention period using a calibrated electronic sphygmomanometer.
16. Echosens Agile 3+ score - composite score comprising LSM, ALT, AST, platelets, age, gender, diabetic status | 6 and 12 months
  Agile 3+ score will be calculated from baseline LSM, ALT, AST, platelets, age, gender and diabetic status and again calculated using the same parameters taken at 26 weeks and at the end of the intervention period.
Health-related Quality of Life assessment - EuroQol EQ-5D-5L to compare the effect of a digital application based lifestyle intervention to standard of care on these | 6 and 12 months
  Health-related Quality of Life will be measured using the EuroQol EQ-5D-5L on day 0, 26 weeks and at the end of the intervention by all participants.
Health-related Quality of Life assessment - Chronic Liver Disease Questionnaire for Nonalcoholic Steatohepatitis (CLDQ-NASH)) - To compare the effect of a digital application based lifestyle intervention to standard of care on these | 6 and 12 months
  Health-related Quality of Life will be measured using the Chronic Liver Disease Questionnaire for Non-alcoholic Steatohepatitis (CLDQ-NASH) on day 0, 26 weeks and at the end of the intervention by all participants.
Hospital Anxiety and Depression Scale (HADS) - To compare the effect of a digital application based lifestyle intervention to standard of care on HADS | 6 and 12 months
  Hospital Anxiety and Depression Scale will be measured on day 0, 26 weeks and at the end of the intervention period by all participants
Number of patients with improvement in liver stiffness measurement LSM - To compare the effect of a digital application based lifestyle intervention to standard of care on number of patients with improvement in LSM | 6 and 12 months
  The total number of patients with improvement in LSM in each group
Liver stiffness measurement - same at primary outcome measure, but at 12 rather than 6 months | 12 months
  The primary outcome measure is change in liver stiffness measurement (LSM) at 6 months compared to baseline. This secondary outcome is that same measure but at 12 months to see if results are sustained. LSM is measured in kPa. VCTE has been validated as a measure of fibrosis across a wide spectrum of chronic liver diseases including MASLD. Whilst liver histology remains the gold standard for fibrosis staging, and magnetic resonance imaging and elastography for non-invasive hepatic lipid quantification and fibrosis respectively, both techniques are largely limited by being time consuming and expensive. VCTE provides multiple advantages of low cost, short procedure time, immediate result availability, good reproducibility and the ability to be performed in an outpatient setting. Studies have shown that LSM has good accuracy for liver-related events and mortality. Change in LSM has been shown to correlate with the risk of liver-related events and death.
Assess the frequency of digital lifestyle application interaction | 12 months
  Gro Health can provide data of individual patient's application usage in the form of total number of 'application openings'. In the intervention group, we would assess whether the participants with more app openings have a greater improvement in their VCTE LSM.
Assess the change in daily step count | 12 months
  In the intervention group, daily step count electronically recorded by compatible smartwatch. Measure mean weekly step count and how this changes over the 12 month period.
Assess the change in amount and type of physical activity | 12 months
  In the intervention group, in addition to daily step count, physical activity can be manually logged by patient (time and date of activity, type of activity and activity duration). Measure weekly total minutes of physical activity and how this changes over the 12 month period.
Assess the change in self-recorded weights | 12 months
  In the intervention group, we would assess the trend in weight loss over the 12 month period
Assess the frequency of food diary usage | 12 months
  In the intervention group, we would assess how frequently participants log food and how this changes over time
Assess the interaction with educational content | 12 months
  Percentage of total educational content reviewed by 12 months. Assess if there is a correlation between amount of educational content reviewed and if this leads to a greater reduction in VCTE LSM.
Number of personalised messages sent to participant over 12 month period | 12 months
  In the intervention group, personalised messages will be sent at least monthly and also ad hoc. We would assess whether the number of messages correlates with change in VCTE LSM.
Total minutes of telephone calls to participant over 12 month period | 12 months
  In the intervention group, telephone calls will be made to participants at 1 week and then ad hoc. We would assess whether the number of minutes correlates with change in VCTE LSM.

CONTACTS AND LOCATIONS:
Locations (1):
- St George's University Hospitals NHS Foundation Trust, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No